CLINICAL TRIAL: NCT04117750
Title: Impact of Vitamin D Supplementation on the Cardiometabolic Status and Androgen Profile in Women With Polycystic Ovary Syndrome: Placebo-Controlled Clinical Trial
Brief Title: Impact of Vitamin D Supplementation on Cardiometabolic Status and Androgen Profile in Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Nearmeen M.Rashad, ass.professor of internal medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: vitamin D and PCO
Record Dates: First submitted 2019-08-27; First posted 2019-10-07 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Evaluations, Diagnostic Self; Treatment Adherence
Keywords: PCOS; VD supplementation; androgen level; cardio metabolic
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Active Comparator): 55 female patients with PCO
  Interventions: Dietary Supplement: cholecalciferol (vit D3)
- non -intervention group (Placebo Comparator): 40 female patients with PCO and 50 healthy women matched to PCOS women as regard age and ethnic origin.
  Interventions: Dietary Supplement: cholecalciferol (vit D3)

INTERVENTIONS:
Dietary Supplement: cholecalciferol (vit D3) — 42,000 IU oral vitamin D per week and 500 mg calcium carbonate
  Other Names: calcium carbonate

SUMMARY:
Polycystic ovary syndrome (PCOS) is a heterogeneous disorder of reproductive, endocrine and metabolic functions. Vitamin D has an influence on metabolic and reproductive functions. This study was designed to explore the levels of free 25 hydroxy cholecalciferol [25(OH) D] in PCOS patients. We also aimed to clarify the impact of vitamin D supplementation on cardiometabolic status, androgen profile and clinical features of PCOS.

DETAILED DESCRIPTION:
Background Polycystic ovarian syndrome (PCOS) is a heterogeneous disorder affecting 510% of women of reproductive age. It is a disorder that affects the reproductive, endocrine and metabolic functions and is the leading cause of chronic anovulation leading to infertility.

PCOS is characterized by hyperandrogenism, chronic oligo or anovulation, and polycystic ovaries. Hyperandrogenism, in particular, is a hallmark feature of PCOS because it is strongly implicated in the genesis of the disorder; and is also associated with metabolic derangements that contribute to the underlying pathophysiology. Also, it is associated with cardiovascular risk factors including obesity, insulin resistance (IR), dyslipidemia, endothelial dysfunction, and metabolic syndrome.

Vitamin D (VD) is a fat-soluble vitamin that is naturally present in very few foods and available as a dietary supplement. It is a steroid hormone with pleiotropic effects. In addition to the main effects of VD on bone and calcium metabolism, it has other roles in the body, including modulation of cell growth, neuromuscular and immune function, and reduction of inflammation.

VD deficiency is now recognized as pandemic disease. Its prevalence varies according to geographic location, season, ethnicity and the standard laboratory value; of what is considered normal, deficient and insufficient. VD deficiency is a risk factor for hypertension, diabetes, and various cancers . Accumulating evidence suggests that VD deficiency might be a causal factor in the pathogenesis of IR and the metabolic syndrome in PCOS. Carotid intima-media thickness (CIMT) measured by ultrasound is a noninvasive, safe, low-cost, reproducible, and well-validated marker of preclinical atherosclerosis.

PCOS is the most frequent endocrine disorder among women of reproductive age and VD deficiency is a key problem in PCOS patients conversely, the basic mechanisms underlying the favorable effects of vitamin D in PCOS are still obscure. Resolving this mechanism may provide insight into the pathophysiology of this syndrome. It can also offer a new therapeutic option for PCOS women. Thus, in the present study was designed to explore the levels of free 25 hydroxyvitamin D [25(OH) D] in PCOS patients. We also aimed to clarify the impact of vitamin D supplementation cardiometabolic status, androgen profile and clinical features of PCOS. Methods This placebo-controlled trial comprised 95 women with PCO recruited from Outpatient Clinics of the Endocrinology Unit of Internal Medicine and Obstetrics and Gynecology Departments, Faculty of Medicine, Zagazig University, Egypt and 50 healthy women matched to PCOS women as regard age and ethnic origin. The diagnosis of PCOS was based on the 2004 revised Rotterdam criteria .. All women underwent the menstrual history and thorough clinical examination. All patients were assessed at the study start on the third day of a spontaneous or progesterone-induced menstrual cycle. Anthropometric measures were estimated, including waist/hip ratio, height and weight then we calculated body mass index (BMI). We estimated the hirsutism score according to Ferriman and Gallwey. .Ovarian volume and antral follicular count (AFC) were evaluated by transvaginal ultrasound (TVS). PCOS patients were randomized divided to the intervention group (n=55) received vitamin D supplements (42,000 IU oral vitamin D per week and 500 mg calcium carbonate per day for 12-week), and non-intervention group (n=40) received 500 mg calcium carbonate per day for 12-week. The exclusion criteria for all women included a history of hyperandrogenic states (such as nonclassic congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome, 21-hydroxylase deficiency, or hyperprolactinemia), DM, hypertension, liver, kidney, or thyroid diseases. In addition, subjects on non-steroidal anti-inflammatory drugs and multivitamin, as well as patients treated with hormone replacement therapy. At the start of the study, the participants were asked to maintain their usual diet and level of physical activity throughout the study period as well as not to receive any lipid-lowering medications and medications that might affect their reproductive physiology during the 12-week intervention. At baseline and at the endpoint of the 12 weeks of study, anthropometrical measurements were estimated as well as and blood samples were collected for biochemical analyses. Written informed consent was taken from all of the participants after explaining details and benefits as well as risks to them. The ethical committee of the Faculty of Medicine, Zagazig University approved our study protocol.

2.1. Sampling of blood Blood samples were drawn from all subjects during the early follicular phase of the menstrual cycles. One ml was collected into tubes containing fluoride for fasting plasma glucose (FPG). A second remaining part underwent immediate serum separation and was stored at -20 ◦C until analysis serum. calcium, phosphate, albumin were measured. Total cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides levels were determined using routine enzymatic methods (Spinreact, Girona, Spain). Low-density lipoprotein (LDL) cholesterol levels were calculated using the Friedewald formula.

2.2. Immunochemical assays: We measured prolactin, FSH, and LH levels via chemiluminescence immunoassays (CLIA) provided by (Immunospec Corporation, CA, USA). Serum high-sensitivity C-reactive protein (hs-CRP) concentrations were measured using high sensitivity enzyme-linked immunosorbent assays (ELISA) (Biosource, Nivelles, Belgium). We determined to fast insulin, FSH, LH, total and free testosterone, sex hormone-binding globulin (SHBG) levels using ELISA kits (DRG International, USA). We calculated insulin resistance (IR) with the homeostatic model assessment (HOMA-IR) index, which is defined as fasting serum insulin (FSI) value (µU/ml) × fasting plasma glucose value (mg/dl)/405. The B cell function was calculated using HOMA- B as (20× (fasting insulin µU/mL)/ (fasting glucose (mmol/l) - 3.5).

2.3.Determination of serum vitamin D levels Serum concentrations of 25(OH)-D were tested using enzyme-linked immunosorbent assay, [Cat No. EQ 6411-9601, Euroimmun Medizinische Labordiagnostika AG, Germany]. Current recommendations define VD deficiency as serum 25(OH)-D levels less than 20 ng/ml and VD insufficiency less than 30 ng/ml.

2.4. Carotid ultrasonography Carotid artery atherosclerosis was determined by one examiner for all patients across all six sites, using high-resolution B-mode ultrasound (M-Turbo®, SonoSite, Washington, Bothell, USA), according to American Society of Echocardiography protocol.

ELIGIBILITY:
Inclusion Criteria:

1. women with PCO. The diagnosis of PCOS was based on the 2004 revised Rotterdam criteria
2. women must be able to swallow tablets

Exclusion Criteria:

1. a history of hyperandrogenic states (such as nonclassic congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome, 21-hydroxylase deficiency, or hyperprolactinemia)
2. DM3-hypertension
3. liver diseases
4. kidney diseases
5. Insulin-dependent diabetes
6. thyroid diseases.
7. women received non-steroidal anti-inflammatory drugs , multivitamins, and hormone replacement therapy.

Ages: 20 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female patient with pco
Enrollment: 145 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
change of lipid profiles in intervention arm of PCOS patients who received vitamin d supplementation | 12 weeks
  change of LDL (mg/dl), TG (mg/dl) TG (mg/dl) ,(mg/dl)
Improvement of fertility ;ovarian size | 12 weeks
  Ovarian volume cm were evaluated by transvaginal ultrasound
change of vitamin D deficiency | 12 weeks
  Serum concentrations of 25(OH)-D( ng/ml )
Change of androgenic levels in intervention arm of PCOS patients who received vitamin d | 12 weeks
  total testosterone (ng/mL),
Change of inflammatory markers in intervention arm of PCOS patients who received vitamin d | 12 weeks
  hs-CRP (µg/ml)
change of BMI | 12 weeks
  weight in kilograms, height in meters
change of fertility , antral follicular count | 12 weeks
  antral follicular count were evaluated by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, El-Shakia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
participants data without names
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after the publication of the study

REFERENCES:
- [Background] Franks S. Polycystic ovary syndrome. N Engl J Med. 1995 Sep 28;333(13):853-61. doi: 10.1056/NEJM199509283331307. No abstract available. PMID 7651477
- [Background] Dunaif A. Insulin resistance and the polycystic ovary syndrome: mechanism and implications for pathogenesis. Endocr Rev. 1997 Dec;18(6):774-800. doi: 10.1210/edrv.18.6.0318. PMID 9408743
- [Background] Lorenz LB, Wild RA. Polycystic ovarian syndrome: an evidence-based approach to evaluation and management of diabetes and cardiovascular risks for today's clinician. Clin Obstet Gynecol. 2007 Mar;50(1):226-43. doi: 10.1097/GRF.0b013e31802f5197. PMID 17304038
- [Background] Talbott E, Guzick D, Clerici A, Berga S, Detre K, Weimer K, Kuller L. Coronary heart disease risk factors in women with polycystic ovary syndrome. Arterioscler Thromb Vasc Biol. 1995 Jul;15(7):821-6. doi: 10.1161/01.atv.15.7.821. PMID 7600112
- [Background] Victor VM, Rocha M, Banuls C, Alvarez A, de Pablo C, Sanchez-Serrano M, Gomez M, Hernandez-Mijares A. Induction of oxidative stress and human leukocyte/endothelial cell interactions in polycystic ovary syndrome patients with insulin resistance. J Clin Endocrinol Metab. 2011 Oct;96(10):3115-22. doi: 10.1210/jc.2011-0651. Epub 2011 Jul 21. PMID 21778215
- [Background] Bikle D. Nonclassic actions of vitamin D. J Clin Endocrinol Metab. 2009 Jan;94(1):26-34. doi: 10.1210/jc.2008-1454. Epub 2008 Oct 14. PMID 18854395
- [Background] Kakarala RR, Chandana SR, Harris SS, Kocharla LP, Dvorin E. Prevalence of vitamin D deficiency in uninsured women. J Gen Intern Med. 2007 Aug;22(8):1180-3. doi: 10.1007/s11606-007-0245-x. Epub 2007 Jun 2. PMID 17546478
- [Background] Hahn S, Haselhorst U, Tan S, Quadbeck B, Schmidt M, Roesler S, Kimmig R, Mann K, Janssen OE. Low serum 25-hydroxyvitamin D concentrations are associated with insulin resistance and obesity in women with polycystic ovary syndrome. Exp Clin Endocrinol Diabetes. 2006 Nov;114(10):577-83. doi: 10.1055/s-2006-948308. PMID 17177140
- [Background] Schmidt-Trucksass A, Grathwohl D, Schmid A, Boragk R, Upmeier C, Keul J, Huonker M. Structural, functional, and hemodynamic changes of the common carotid artery with age in male subjects. Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):1091-7. doi: 10.1161/01.atv.19.4.1091. PMID 10195940
- [Background] Bianchini E, Bozec E, Gemignani V, Faita F, Giannarelli C, Ghiadoni L, Demi M, Boutouyrie P, Laurent S. Assessment of carotid stiffness and intima-media thickness from ultrasound data: comparison between two methods. J Ultrasound Med. 2010 Aug;29(8):1169-75. doi: 10.7863/jum.2010.29.8.1169. PMID 20660450
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] FERRIMAN D, GALLWEY JD. Clinical assessment of body hair growth in women. J Clin Endocrinol Metab. 1961 Nov;21:1440-7. doi: 10.1210/jcem-21-11-1440. No abstract available. PMID 13892577
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Stein JH, Korcarz CE, Hurst RT, Lonn E, Kendall CB, Mohler ER, Najjar SS, Rembold CM, Post WS; American Society of Echocardiography Carotid Intima-Media Thickness Task Force. Use of carotid ultrasound to identify subclinical vascular disease and evaluate cardiovascular disease risk: a consensus statement from the American Society of Echocardiography Carotid Intima-Media Thickness Task Force. Endorsed by the Society for Vascular Medicine. J Am Soc Echocardiogr. 2008 Feb;21(2):93-111; quiz 189-90. doi: 10.1016/j.echo.2007.11.011. No abstract available. PMID 18261694